CLINICAL TRIAL: NCT04071184
Title: Phase 1b Clinical Study of the Safety and Pharmacokinetics of Alofanib in Patients With Metastatic Gastric Cancer Resistant to Standard Therapy
Brief Title: Study of Alofanib in Patients With Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Pharmaceutical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPT835GC1B
Record Dates: First submitted 2019-08-13; First posted 2019-08-28 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; metastases; patients with previous treatment failures; FGFR2 abnormalities
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — alofanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose cohorts (Experimental): Part 1 (dose escalation): "3+3" design will be used. Alofanib (dose levels of 50, 100, 165, 250, 350 mg/m2) will be given i.v. daily (1-5 days on, 6-7 days off, every week) till progression or unacceptable toxicity.
  Part 2 (dose expansion): Afterwards the dosing regimen identified in Part 1 will be evaluated in a single-arm study focused on clinical efficacy.
  Interventions: Drug: Alofanib

INTERVENTIONS:
Drug: Alofanib — Five dose cohorts and expanded cohort will be included

SUMMARY:
This is a non-randomized multicenter phase 1b clinical trial of the safety and pharmacokinetics, as well as the preliminary efficacy of monotherapy with alofanib, an allosteric fibroblast growth factor receptor 2 inhibitor, in patients with advanced gastric cancer who have exhausted the resource of standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric cancer (adenocarcinoma)
* Progression of the disease (clinical and/or radiological) on previous standard systemic therapy
* Measurable lesions according to the RECIST 1.1 criteria
* Possibility to assess the amplification of FGFR2, fusion of FGFR2 genes, overexpression of FGFR2, phosphorylation of FRS2
* ECOG PS 0-2
* Age >= 18 years old
* Adequate function of organs
* Absence of any psychological, family, social or geographical circumstances that could potentially serve as obstacles to the implementation of the study
* Patients capable of childbearing should use an effective method of contraception
* Signed Informed Consent

Exclusion Criteria:

* Participation in another clinical study and concomitant treatment with any research drug or any study of antitumor therapy, including radiation, within 28 days before inclusion in this study
* Presence of metastases in the central nervous system and / or carcinoma of the meninges at the time of inclusion in the study
* Presence or history of present signs of any condition, therapy or laboratory abnormalities that could limit the interpretation of the results of this study
* Any malignant tumor within the previous 5 years, with the exception of adequately cured cervical cancer in situ or squamous cell skin cancer, or basal cell skin cancer with limited growth, subject to adequate control over the course of this disease
* Pregnancy
* Known positive status for human immunodeficiency virus (HIV) or active hapatitis B and C
* Surgery within 7 days before the first dose of the study drug
* Signs of bleeding or hemorrhagic diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-26 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or Recommended phase 2 dose (RP2D) | 6 months
  The highest dose of an alofanib that does not cause unacceptable side effects and recommended

SECONDARY OUTCOMES:
Cmax | 1 month
  Peak Plasma Concentration (Cmax), the maximum concentration recorded
Tmax | 1 month
  Time of Maximum concentration observed
AUC | 1 month
  Area under the plasma concentration versus time curve
t1/2 | 1 month
  Elimination half-life, the time taken for the plasma concentration to fall by half its original value
CL | 1 month
  blood clearance
Vd | 1 month
  Volume of distribution, the theoretical volume that would be necessary to contain the total amount of an alofanib at the same concentration that it is observed in the plasma
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | 12 months
  Rate of AEs and SAEs according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Progression-free survival (PFS) | 12 months
  PFS is defined as the time from treatment start to disease progression or death from any cause
Overall survival (OS) | 12 months
  OS is defined as the time from treatment start to death from any cause
Objective response rate (ORR) | 12 months
  ORR is the proportion of patients with tumor size reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Tsimafeyeu, MD, Study Director — Scientific Adviser
Locations (4):
- Russia (4):
  - N.N.Blokhin Russian Cancer Research Centre, Dept. of Clinical Pharmacology and Chemotherapy, Moscow
  - Omsk Regional Cancer Center, Omsk
  - Rostov Research Institute of Oncology, Rostov-on-Don
  - St. Petersburg City Cancer Center, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsimafeyeu I, Statsenko G, Vladimirova L, Besova N, Artamonova E, Raskin G, Rykov I, Mochalova A, Utyashev I, Gorbacheva S, Kazey V, Gavrilova E, Dragun N, Moiseyenko V, Tjulandin S. A phase 1b study of the allosteric extracellular FGFR2 inhibitor alofanib in patients with pretreated advanced gastric cancer. Invest New Drugs. 2023 Apr;41(2):324-332. doi: 10.1007/s10637-023-01340-z. Epub 2023 Mar 13. PMID 36907947